CLINICAL TRIAL: NCT07221591
Title: Relative Bioavailability of Two Survodutide (BI 456906) Formulations When Administered Subcutaneously Via Pre-filled Syringe Over 28 Weeks (an Open-label, Randomised, Multiple Dose, Parallel Group Trial)
Brief Title: A Study in Healthy People to Compare How 2 Different Formulations of Survodutide Are Taken up by the Body
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0103; 2025-522325-35-00 (EU CTIS Number); U1111-1322-4700 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-10-27; First posted 2025-10-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- survodutide formulation A (reference treatment) (Active Comparator)
  Interventions: Drug: survodutide
- survodutide formulation B2 (test treatment) (Experimental)
  Interventions: Drug: survodutide

INTERVENTIONS:
Drug: survodutide — survodutide

SUMMARY:
This study is open to healthy people between 18 and 65 years of age. People can join the study if they have a body mass index between 27 and 39.9 kg/m2.

The purpose of this study is to test a new formulation of a medicine called survodutide. Survodutide is being developed to help people with obesity and people with liver conditions. When a new formulation is developed, it is important to understand how it is taken up by the body.

Participants are divided into 2 groups by chance. One group gets the reference formulation of survodutide (formulation A). The other group gets the new formulation of survodutide (formulation B2). Participants in both groups inject survodutide under their skin once a week for about 6 and a half months.

Participants are in the study for about 7 months. During this time, they visit the study site 15 times. For one of the visits, participants stay overnight for 3 nights at the study site. The site staff takes blood samples to measure how much survodutide is in the blood. They also check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

* Healthy male or female trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* Body mass index (BMI) of 27.0 to 39.9 kg/m² (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial Further inclusion criteria apply.

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 150 mmHg, diastolic blood pressure outside the range of 50 to 100 mmHg, or pulse rate outside the range of 50 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator. Presence of hypertension, hypothyroidism, hyperuricaemia and hypercholesterolaemia are acceptable if well-controlled according to the investigator's judgement.

Further exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | up to 232 days
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | up to 232 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - CRS Clinical Research Services Mannheim GmbH, Mannheim

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com